CLINICAL TRIAL: NCT01918176
Title: A Phase 1, Open-Label Fixed-Sequence 2-Period Crossover Study Of Palbociclib In Healthy Subjects To Investigate The Potential Effect Of Antacid Treatment On The Pharmacokinetics Of A Single Oral Dose Administered Under Fasted Conditions
Brief Title: Drug Interaction Study To Investigate The Potential Effect Of Proton Pump Inhibitor On The Pharmacokinetics Of Palbociclib (PD-0332991)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A5481018
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Healthy
Keywords: Palbociclib; PD-0332991; Proton Pump Inhibitor; DDI; Healthy Volunteers; Pharmacokinetics; Rabeprazole
MeSH Terms: interventions — palbociclib; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fixed sequence crossover (Experimental): All the subjects will undergo the treatment of Palbociclib alone first and then treatment of Palbociclib and Rabeprazole.
  Interventions: Drug: Palbociclib alone; Drug: Palbociclib + Rabeprazole

INTERVENTIONS:
Drug: Palbociclib alone — Single dose of 125mg Palbociclib capsule will be administered to subjects orally and then PK samples will be collected at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours.
  Other Names: Period 1
Drug: Palbociclib + Rabeprazole — Two Rabeprazole 20mg tablets will be given to subjects orally once daily for 7 days. Then on the same day at least 4 hours after the last dose of Rabeprazole, single dose of 125mg Palbociclib capsule will be given to subjects orally then followed by PK samplings at 1, 2, 4, 6, 8, 12, 24, 48, 72, 96 and 120 hours.
  Other Names: Period 2

SUMMARY:
Fixed sequence, 2-period crossover study to compare the pharmacokinetic profiles of Palbociclib in absence and presence of prior administration of proton pump inhibitor Rabeprazole. The increased gastric pH achieved by the treatment with multiple doses of Rabeprazole might affect the absorption process of Palbociclib.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects of non-childbearing potential; Healthy subjects identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory test.

Exclusion Criteria:

* A positive urine drug screen, urine cotinine test or alcohol breath test.
* Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives prior to the first dose of study medication. All antacid agents must be discontinued 28 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 0-120 hours
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 0-120 hours

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] | 0-120 hours
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Area Under the Curve from Time Zero to 72 hours | 0-72 hours
  AUC (0-t)= Area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hours
Apparent Oral Clearance (CL/F) | 0-120 hours
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0-120 hours
Time For the Last Quantifiable Concentration (Tlast) | 0-120 hours
Apparent Volume of Distribution (Vz/F) | 0-120 hours
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Plasma Decay Half-Life (t1/2) | 0-120 hours
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481018